CLINICAL TRIAL: NCT00534144
Title: A Randomized Controlled Trial of the Effect of IV Iron on Proteinuria in Non-Dialysis Chronic Kidney Disease Patients
Brief Title: Comparison Between Effects of Two Iron Preparations on Protein in the Urine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FER0701
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Failure, Chronic; Anemia, Iron-Deficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; ferric gluconate; Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron Sucrose (Active Comparator)
  Interventions: Drug: iron sucrose injection, USP
- Ferric Gluconate (Active Comparator)
  Interventions: Drug: sodium ferric gluconate complex in sucrose injection

INTERVENTIONS:
Drug: iron sucrose injection, USP — iron sucrose injection, USP, 100 mg intravenously (IV) per week, for 5 weeks
  Arms: Iron Sucrose
Drug: sodium ferric gluconate complex in sucrose injection — sodium ferric gluconate complex in sucrose injection, 100 mg intravenously (IV) per week, for 5 weeks
  Arms: Ferric Gluconate

SUMMARY:
This study will compare the effects of sodium ferric gluconate complex and iron sucrose on urine concentrations of various chemicals including protein

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe anemia
* Iron deficiency
* Moderate to severe chronic kidney disease, not receiving dialysis
* Age ≥ 18 or greater and able to give informed consent

Exclusion Criteria:

* Known sensitivity to Sodium Ferric Gluconate Complex in Sucrose Injection, Iron sucrose USP, or any of their components
* Clinically unstable
* Indication of iron sufficiency
* Bladder obstruction conditions that would not allow for good urine output

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in urine protein | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naomi V. Dahl, Pharm.D., Study Director — Watson Laboratories, Inc.
Locations (13):
- United States (12):
  - Phoenix, Arizona
  - Alhambra, California
  - Bell Gardens, California
  - Exeter, California
  - Glendale, California
  - Visalia, California
  - Fort Lauderdale, Florida
  - Hines, Illinois
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Houston, Texas
  - Fairfax, Virginia
- San Juan, Puerto Rico

REFERENCES:
- [Result] Agarwal R, Leehey DJ, Olsen SM, Dahl NV. Proteinuria induced by parenteral iron in chronic kidney disease--a comparative randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jan;6(1):114-21. doi: 10.2215/CJN.06020710. Epub 2010 Sep 28. PMID 20876669